CLINICAL TRIAL: NCT00153543
Title: Immunogenicity and Reactogenicity of Pneumococcal Polysaccharide and Conjugate Vaccines in Native Elders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Alaska Native Tribal Health Consortium (Other); Southcentral Foundation (Other)
Responsible Party: Principal Investigator, Karen Miernyk, Laboratory Manager, Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCID-3316
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections

ARMS (3):
- PPV23 (Active Comparator): Receive one dose of PPV23
  Interventions: Biological: PCV7 + PPV23, 2 months; Biological: PCV7 + PPV23, 6 months
- PCV7 + PPV23, 2 months (Experimental): Receive one dose of PCV7 + 1 dose of PPV23 2 months later
  Interventions: Biological: PCV7 + PPV23, 6 months
- PCV7 + PPV23, 6 months (Experimental): Receive one dose of PCV7 + 1 dose of PPV23 6 months later
  Interventions: Biological: PCV7 + PPV23, 2 months

INTERVENTIONS:
Biological: PCV7 + PPV23, 2 months
  Arms: PCV7 + PPV23, 6 months; PPV23
Biological: PCV7 + PPV23, 6 months
  Arms: PCV7 + PPV23, 2 months; PPV23

SUMMARY:
To test the hypothesis that immune responses to 23-valent pneumococcal polysaccharide vaccine (PPV-23) could be improved in Alaska Native elders by immune priming with 7-valent pneumococcal conjugate vaccine (PCV-7), we assessed post-vaccination immune responses among Natives aged 55 years and older who were randomized into three arms: (1) one dose of PPV-23 according to current state and ACIP recommendations; (2) one dose of PCV-7 followed two months later with a dose of PPV-23; and (3) one dose of PCV-7 followed six months later with a dose of PPV-23.

DETAILED DESCRIPTION:
Rates of invasive pneumococcal infection (bacteremia and meningitis caused by Streptococcus pneumoniae) for Alaska Natives are among the highest in the United States and are approximately five-fold higher than rates among non-Natives living in Alaska. Disease is most common among the very young and the elderly (73 cases/100,000 Natives ≥55 years old)1. Case-fatality from pneumococcal infection is highest (>15%) among the elderly. A 23-valent pneumococcal polysaccharide vaccine (PPV-23) has been licensed in the United States since 1983. The CDC Advisory Committee on Immunization Practices (ACIP) recommends vaccination with PPV-23 for all Alaska Natives aged two years and older, however the Alaska Department of Health and the Alaska Native Tribal Health Consortium only target and fund vaccination for those aged 55 years and older. Post-licensure epidemiological studies have documented effectiveness of PPV-23 for prevention of invasive infection (bacteremia and meningitis) among the elderly and younger adults with certain chronic medical conditions. The overall effectiveness against invasive pneumococcal disease among immunocompetent persons age ≥65 years is 75%; however, efficacy may decrease with advancing age.

PPV-23 has several limitations. Efficacy of pneumococcal polysaccharide vaccines against the most common types of pneumococcal infection in the elderly, bronchitis and pneumonia without bacteremia, has not been documented in controlled, randomized trials. Additionally, antibodies against pneumococcal polysaccharides decline after immunization and often return to pre-vaccination concentrations within 5 years. A case-control study evaluating vaccine effectiveness suggests that the decline in antibody concentration is associated with declining protection against invasive pneumococcal infection. At present, the Alaska Department of Health recommends revaccination with PPV-23 every 6 years. This is in contrast to ACIP recommendations for only one revaccination. A retrospective review found similar rates of local and systemic reactions among 179 Alaska Native elders who received a third dose of PPV-23 compared to 180 receiving a first or second dose. Although available data suggest that revaccination with PPV-23 is safe, clinical benefits of revaccination are unproven. T-cell independent antigens, such as polysaccharides, do not produce booster responses to revaccination, and antibody levels after revaccination do not exceed those after primary immunization.

A 7-valent pneumococcal conjugate vaccine (PCV-7) was licensed in 2000 (Prevnar™, Wyeth Lederle Vaccines) for prevention of invasive pneumococcal disease in infants and young children. This vaccine was safe and effective for prevention of invasive pneumococcal disease in a large randomized trial conducted among infants aged two months and older enrolled in a northern California HMO. The role of pneumococcal conjugate vaccines among adults has not been defined. Potential advantages of conjugate vaccines compared to PPV-23 include the T-cell dependent immune response to conjugate vaccines which lead to immunologic memory and booster responses characterized by rapid and dramatic increases in antibody after revaccination. PCV-7 should also overcome the limitations of the poorly immunogenic antigens in PPV-23, including those resistant to antimicrobial drugs. An additional potential advantage of PCV-7 is greater mucosal immunity with possible protection against non-bacteremic pneumococcal respiratory tract infections-a benefit that has never been confirmed for PPV-23 among the elderly. Potential disadvantages of PCV-7 in adults include limited serotype coverage. Only 50% of invasive pneumococcal infections in Alaska Natives aged 55 and older are caused by the seven serotypes included in PCV-7 compared to more than 90% for PPV-23. Preliminary data from studies of healthy persons ≥50 years old and of patients vaccinated after treatment for Hodgkin's disease indicate that antibody responses to a dose of pneumococcal conjugate vaccine have not been substantially better than responses to PPV-23. One approach to the use of conjugate vaccines in adults is to administer conjugate vaccine to prime the immune system and to subsequently give a dose of PPV-23 to induce a booster response to the serotypes present in both vaccines as well as primary T-cell independent responses to the serotypes in PPV-23 only. Immunogenicity studies have documented boosting with polysaccharide vaccine in children with chronic illnesses and in adults with Hodgkin's Disease after primary vaccination with pneumococcal conjugate vaccine. However, there are no published data evaluating this strategy for preventing pneumococcal disease in the elderly, and no data are available for Alaska Natives.

We studied the immunogenicity of PCV-7 in Alaska Native elders. Participants were randomized into three arms: (1) one dose of PPV-23 according to current state and ACIP recommendations; (2) one dose of PCV-7 followed two months later with a dose of PPV-23; and (3) one dose of PCV-7 followed six months later with a dose of PPV-23. Immune responses for all conjugate vaccine pneumococcal serotypes will be determined by enzyme linked immunosorbent assay (ELISA) and antibody affinity at the Centers for Disease Control and Prevention's (CDC) Arctic Investigations Program (AIP) laboratory located on the Alaska Native Medical Center (ANMC) campus.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 to 70 years
* Alaska Native

Exclusion Criteria:

* Immune compromising condition
* Neurological disease
* Immune suppressive medication or immunoglobulin within 6 months
* Previous pneumococcal vaccination

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2002-05 (Actual); Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Miernyk, MS, Principal Investigator — Alaska Native Tribal Health Consortium
Locations (1):
- Alaska Native Medical Center, Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data can be shared.

REFERENCES:
- [Result] Miernyk KM, Butler JC, Bulkow LR, Singleton RJ, Hennessy TW, Dentinger CM, Peters HV, Knutsen B, Hickel J, Parkinson AJ. Immunogenicity and reactogenicity of pneumococcal polysaccharide and conjugate vaccines in alaska native adults 55-70 years of age. Clin Infect Dis. 2009 Jul 15;49(2):241-8. doi: 10.1086/599824. PMID 19522655

RESULTS

PARTICIPANT FLOW:
Groups:
- PPV23: Receive one dose of PPV23
  PCV7 + PPV23, 2 months
  PCV7 + PPV23, 6 months
- PCV7 + PPV23, 2 Months: Receive one dose of PCV7 + 1 dose of PPV23 2 months later
  PCV7 + PPV23, 6 months
- PCV7 + PPV23, 6 Months: Receive one dose of PCV7 + 1 dose of PPV23 6 months later
  PCV7 + PPV23, 2 months
Period: Overall Study
Arm/Group | PPV23 | PCV7 + PPV23, 2 Months | PCV7 + PPV23, 6 Months
Started | 28 | 29 | 29
Completed | 28 | 29 | 27
Not Completed | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PPV23 | PCV7 + PPV23, 2 Months | PCV7 + PPV23, 6 Months | Total
Number analyzed (Participants) | 28 | 29 | 29 | 86
Age, Continuous [Median (Full Range); unit: years] | 57 [55 to 66] | 58 [55 to 66] | 58 [55 to 69] | 58 [55 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 17 | 52
  Male | 10 | 12 | 12 | 34
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 29 | 29 | 86
Anti-pneumococcal antibody concentrations [Geometric Mean (Full Range); unit: ug/mL]
  serotype 1 | 0.35 [0.21 to 0.58] | 0.39 [0.23 to 0.64] | .40 [.21 to .73] | 0.38 [0.21 to 0.73]
  serotype 4 | .14 [.08 to .25] | .22 [.14 to .36] | .17 [.1 to .29] | 0.18 [0.08 to 0.36]
  serotype 6B | 1.57 [.93 to 2.65] | 1.72 [1.14 to 2.58] | 1.67 [1.09 to 2.54] | 1.65 [0.93 to 2.65]
  serotype 14 | 2.61 [1.35 to 5.07] | 2.32 [1.17 to 4.59] | 1.9 [1.08 to 3.32] | 2.28 [1.08 to 5.07]
  serotype 19F | 2.36 [1.6 to 3.49] | 2.34 [1.61 to 3.39] | 1.8 [1.2 to 2.72] | 2.17 [1.2 to 3.49]

OUTCOME MEASURES:

1. Primary Outcome: Immune Responses
Description: antibody titers to 5 pneumococcal serotypes
Time Frame: 2 months after final dose of vaccine
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | PPV23 | PCV7 + PPV23, 2 Months | PCV7 + PPV23, 6 Months
Number analyzed (Participants) | 28 | 29 | 27
ug/mL
  serotype 1 | 1.95 [1.21 to 3.15] | 1.69 [1.03 to 2.76] | 1.22 [0.59 to 2.52]
  serotype 4 | 0.78 [.43 to 1.42] | 1.23 [.77 to 1.97] | .8 [.52 to 1.23]
  serotype 6B | 4.1 [2.33 to 7.19] | 4.22 [2.45 to 7.29] | 5.05 [2.63 to 9.71]
  serotype 14 | 6.62 [3.58 to 12.24] | 6.82 [3.31 to 14.07] | 11.13 [6.26 to 19.82]
  serotype 19F | 5.05 [3.3 to 7.74] | 6.62 [4.4 to 9.95] | 8.1 [6.22 to 12.53]

2. Secondary Outcome: Number of Participants With Systemic and Injection Site Reactions
Description: Systemic and local injection site reactions as measured by participants with follow up with study staff
Time Frame: every day for 3 days after each injection
Measure: Count of Participants; unit: Participants
Arm/Group | PPV23 | PCV7 + PPV23, 2 Months | PCV7 + PPV23, 6 Months
Number analyzed (Participants) | 28 | 29 | 29
Participants
  any redness at injection site | 2 | 10 | 7
  any swelling at injection site | 6 | 20 | 17
  any arm pain in injected arm | 20 | 26 | 27
  All-cause mortality | 0 | 0 | 0
  Serious adverse events | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | PPV23 | PCV7 + PPV23, 2 Months | PCV7 + PPV23, 6 Months
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 20/28 | 26/29 | 27/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PPV23 (N=28) | PCV7 + PPV23, 2 Months (N=29) | PCV7 + PPV23, 6 Months (N=29)
any arm pain in injected arm (General disorders) | 20 (20) | 26 (26) | 27 (27) — pain in the subject's arm where they received the vaccine injection
any redness at injection site (General disorders) | 2 (2) | 10 (10) | 7 (7) — redness in the subject's arm where they received the vaccine injection
any swelling at injection site (General disorders) | 6 (6) | 20 (20) | 17 (17) — swelling in the subject's arm where they received the vaccine injection

LIMITATIONS AND CAVEATS:
There were a small number of subjects in each study group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No